CLINICAL TRIAL: NCT06466564
Title: A Prospective, Multi-center, Open-label, Non-inferiority, Randomized, Controlled Trial of Bioabsorbable/Nufairy Coil Embolization System for the Treatment of Intracranial Aneurysms
Brief Title: Bioabsorbable/Nufairy Coil Application Trial in China
Acronym: NuCATCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSTH-2023-02-0A
Record Dates: First submitted 2024-03-04; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Bioabsorbable/Nufairy coil embolization system
  Interventions: Device: Nufairy® Coil embolization system for intracranial aneurysm
- Control group (Active Comparator): Numen coil embolization system
  Interventions: Device: Nufairy® Coil embolization system for intracranial aneurysm

INTERVENTIONS:
Device: Nufairy® Coil embolization system for intracranial aneurysm — Nufairy® Coil embolization system for intracranial aneurysm

SUMMARY:
The scope of this trial is the collection and analysis of effectiveness and safety endpoints, related to the use of the Bioabsorbable/Nufairy Coil Embolization System in the treatment of intracranial aneurysms.

DETAILED DESCRIPTION:
Approximately 258 subjects with intracranial aneurysms would be enrolled for coiling embolization according to the inclusion and exclusion criteria specified in this trial protocol. Subjects were evaluated by mRS preoperatively, at the time of device implantation, at the time of discharge from the hospital, at 1 month (±7 days) postoperatively, at 6 months (±30 days) postoperatively, and at 12 months (±90 days) postoperatively; subjects would underwent DSA imaging at surgery and at 12months (±90 days) postoperatively, and MRA imaging at 18 months (±90 days) postoperatively. Unplanned follow-up of the subjects would performed when necessary, and data would be recorded to evaluate the safety and efficacy of Nufairy Coil Embolization System for coiling embolization for the treatment of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old and ≤80 years old at the time of signing the informed consent;
2. Intracranial aneurysm diagnosed by CTA, MRA, DSA neuroimaging examination;
3. Subjects whose target aneurysms are suitable for embolization with flow diverter or intracranial arterial stents assisted by coils, and the entire treatment can be performed in a single procedure;
4. The subjects or the subject's guardian signs the informed consent voluntarily and is willing to accept follow-up.

Exclusion Criteria:

1. mRS Score ≥3 points in clinical assessment prior to enrollment;
2. Subjects who received neurosurgical or endovascular treatment for recurrent aneurysms;
3. Subjects with multiple aneurysms;
4. Subjects with ruptured aneurysms <30 days;
5. Significant stenosis (≥50%) of parent artery;
6. Subjects who are not suitable for anesthesia or intravascular surgery, such as major diseases of the heart, lung, liver, spleen, kidney, brain tumors, severe active infections, disseminated intravascular coagulation, and a history of serious mental illness;
7. Subjects who have undergone major surgical procedures (such as internal fixation device implantation of limbs fracture, tumor resection, major organ surgery, etc.) within 30 days before signing the informed consent or plan to undergo major surgical procedures within 60 days after signing the informed consent;
8. Subjects with morphology or lesions that may interfere with device use, including but not limited to: carotid artery dissection, vasculitis, aortic dissection, limited vascular access (e.g., severe intracranial vessel tortuosity, severe intracranial vessel spasm that does not respond to medical treatment, other anatomical or clinical changes that impede device access;
9. Treatment contrainidations of coils, including but not limited to: contrainidations of digital subtraction angiography, allergy to or intolerance of contrast agents, allergy to or intolerance of anti-platelet and anticoagulant drugs required for treatment, platinum-tungsten alloy, and poly(co-glycolic acid) (PLGA);
10. Pregnant or lactating women;
11. Life expectancy is less than 18 months;
12. Subjects participating in other drug or device studies did not meet the endpoint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-12-24 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Successful occlusion rate of aneurysm at 12-month post-procedure. | 12 month
  It was defined as the percentage of subjects with the degree of aneurysm embolization scored as Raymond I or II (i.e., 95%-100% aneurysm embolization).

SECONDARY OUTCOMES:
Complete occlusion rate of aneurysm at 12-month post-procedure. | 12 month
  The "complete occlusion rate of aneurysm" was defined as the percentage of subjects with the degree of aneurysm embolization scored as Raymond I (i.e., 100% aneurysm embolization).
Recurrence rate of aneurysm at 12-month post-procedure. | 12 month
  The "recurrence rate of aneurysm" was defined as the percentage of subjects with a decrease in the degree of aneurysm embolization at the follow-up visit as compared with immediately post-procedure.
Retreatment rate of aneurysm at 12-month post-procedure. | 12 month
  The "retreatment of aneurysm" was defined as the percentage of subject who received retreatment for the recurrence of target aneurysms during the follow-up period
Device-related serious adverse events at 1, 6, and 12 months after surgery; | 12 month
The incidence of ipsilateral stroke or neurologic death of the target aneurysm within 12 months. | 12 month
The incidence of ipsilateral ischemic stroke of the target aneurysm within 12 months. | 12 month

OTHER OUTCOMES:
Successful occlusion rate of aneurysm at 18-month post-procedure. | 18 month
  It was defined as the percentage of subjects with the degree of aneurysm embolization scored as Raymond I or II (i.e., 95%-100% aneurysm embolization).
Recurrence rate of aneurysm at 18-month post-procedure. | 18 month
  The "recurrence rate of aneurysm" was defined as the percentage of subjects with a decrease in the degree of aneurysm embolization at the follow-up visit as compared with immediately post-procedure.
Retreatment rate of aneurysm at 18-month post-procedure. | 18 month
  The "retreatment of aneurysm" was defined as the percentage of subject who received retreatment for the recurrence of target aneurysms during the follow-up period
The incidence of ipsilateral stroke or neurologic death of the target aneurysm within 18 months. | 18 month
Device-related serious adverse events at 18 months after surgery | 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China